CLINICAL TRIAL: NCT07233577
Title: The Effect of Dexamethasone in Full Pulpotomy on Postoperative Pain in Permanent Molars With Symptomatic Irreversible Pulpitis: A Randomized Clinical Study
Brief Title: The Effect of Dexamethasone in Full Pulpotomy on Postoperative Pain in Permanent Molars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Kübra Gürler, Principal Investigator, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 06.12.2024/15
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Pulpitis - Irreversible
MeSH Terms: interventions — Cryotherapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): The pulp chamber was irrigated with 5 mL of sterile saline at room temperature (22-25°C). The solution was delivered slowly into the pulp chamber using a sterile syringe with a blunt needle tip and left in place for 5 minutes to allow direct contact with the exposed radicular pulp tissue. Afterward, the chamber was dried gently with sterile cotton pellets.
- Cryotherapy Group (Experimental): 5 mL of sterile saline solution pre-cooled to 2.5°C was administered into the pulp chamber using the same technique. This solution was also left in contact with the pulp tissue for 5 minutes, without aspiration, to provide localized cold exposure. The cold saline was stored in a calibrated medical cooler and monitored with a digital thermometer to ensure consistent temperature throughout the clinical procedure.
  Interventions: Other: Cryotherapy
- Dexamethasone Group (Experimental): The pulp chamber was irrigated with 2 mL of a dexamethasone sodium phosphate solution at a concentration of 4 mg/mL (Decort®, DEVA Holding, Türkiye). The solution was slowly delivered into the pulp chamber using a sterile syringe with a blunt-tipped needle and left in place for 1 minute to allow direct contact with the exposed radicular pulp tissue. Subsequently, the chamber was gently dried with sterile cotton pellets.
  Interventions: Drug: Dexametasone

INTERVENTIONS:
Other: Cryotherapy — In the cryotherapy group, the pulp chamber was irrigated with 5 mL of sterile saline solution pre-cooled to 2.5°C during full pulpotomy.
  Arms: Cryotherapy Group
Drug: Dexametasone — In the dexamethasone group, the pulp chamber was irrigated with 2 mL of dexamethasone sodium phosphate solution (4 mg/mL) during full pulpotomy.
  Arms: Dexamethasone Group

SUMMARY:
The goal of this clinical trial is to evaluate the effects of cryotherapy and dexamethasone on the intensity of postoperative pain in full pulpotomy procedures in permanent molars with symptomatic irreversible pulpitis. The main questions it aims to answer are:

* Does controlled irrigation with cold saline during full pulpotomy reduce the severity of postoperative pain?
* Does controlled irrigation with dexamethasone during full pulpotomy reduce the severity of postoperative pain? In the cryotherapy group, unlike the control and dexamethasone groups, the pulp chamber was irrigated with 2°C saline solution during the final irrigation step.

In the dexamethasone group, unlike the control and cryotherapy groups, the pulp chamber was irrigated with 2 mL dexamethasone solution during the final irrigation step.

ELIGIBILITY:
Inclusion Criteria:

* Vital permanent molars exhibiting positive responses to both the cold test and the electric pulp test, with a prolonged cold response (>30 seconds) consistent with symptomatic irreversible pulpitis.
* Presence of deep carious lesions in the included teeth (indicated for vital pulp therapy).
* No radiographic evidence of periapical pathology (i.e., no periapical radiolucency, root resorption, or pathological widening of the periodontal ligament space).
* Patients who had not taken analgesics or antibiotics during the 24 hours preceding the procedure.

Exclusion Criteria:

* Devital permanent molars that responded negatively to cold tests and electric pulp tests
* Permanent molars with poor periodontal status (pocket depth > 4 mm),
* Teeth that exhibited periapical radiolucency, pathological mobility, or were deemed non-restorable
* Systemic diseases, pregnancy or lactation, known allergies to dexamethasone or NSAIDs, recent use of analgesics (within 24 hours), and any contraindications for pulpotomy or local anesthesia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2024-12-18 (Actual); Primary Completion 2025-05-05 (Actual); Study Completion 2025-06-16 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | up to 72 hours
  The visual analog scale for pain is a straight line with one end meaning no pain (0) and the other end meaning the worst pain (10) imaginable. A patient marks a point on the line that matches the amount of pain he or she feels. It may be used to help choose the right dose of pain medicine. Also called VAS.

CONTACTS AND LOCATIONS:
Overall Officials: Koray Yılmaz, DDS, MSc, Professor, Principal Investigator — Cukurova University
Locations (1):
- Cukurova University, Adana, Sarıçam, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dildar I, Moghal A, Mirza A, Zaheer MA, Mallick MR, Munir S. Evaluation of Postoperative Pain after Using Dexamethasone Intracanal Rinse in Irreversible Pulpitis. J Coll Physicians Surg Pak. 2024 Apr;34(4):390-393. doi: 10.29271/jcpsp.2024.04.390. PMID 38576278
- [Background] Solomon RV, Paneeru SP, Swetha C, Yatham R. Comparative evaluation of effect of intracanal cryotherapy and corticosteroid solution on post endodontic pain in single visit root canal treatment. J Clin Exp Dent. 2024 Mar 1;16(3):e250-e256. doi: 10.4317/jced.61023. eCollection 2024 Mar. PMID 38600937
- [Background] Rogers MJ, Johnson BR, Remeikis NA, BeGole EA. Comparison of effect of intracanal use of ketorolac tromethamine and dexamethasone with oral ibuprofen on post treatment endodontic pain. J Endod. 1999 May;25(5):381-4. doi: 10.1016/S0099-2399(06)81176-3. PMID 10530266